CLINICAL TRIAL: NCT07203378
Title: ENERGIZE: Engagement With a Nurturing Exercise Routine for Greater Improvement in Zest and Energy on Enhertu: A Single-Center Pilot Study
Brief Title: Nurturing Exercise Routine for Greater Improvement in Zest and Energy on Enhertu
Acronym: ENERGIZE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCI194215
Record Dates: First submitted 2025-09-17; First posted 2025-10-02 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-09

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Intervention (Experimental)
  Interventions: Other: Whole-body resistance training and aerobic exercise
- Usual Care (No Intervention)

INTERVENTIONS:
Other: Whole-body resistance training and aerobic exercise — A 12-week individualized, home-based, unsupervised, whole-body resistance training and aerobic exercise routine will be provided to each study participant.
  Arms: Exercise Intervention

SUMMARY:
The goal of this study is to test the efficacy of using a 12-week, home-based, unsupervised aerobic and resistance training exercise program for changes in cancer-related fatigue in patients with metastatic breast cancer who are receiving Enhertu.

ELIGIBILITY:
Inclusion Criteria:

* Subject aged ≥ 18 years
* Diagnosis of locally advanced/unresectable or metastatic breast cancer.
* Has received 3 or 4 cycles of Enhertu and is expected to continue treatment for at least 12 weeks.
* Able and willing to participate in the interventional aerobic exercise and resistance exercises.
* Currently following standard of care contraception requirements and willing to continue following these requirements for the duration of therapy.
* Able to provide informed consent and willing to sign an approved consent form that conforms to federal and institutional guidelines.
* Experiencing clinical fatigue symptoms in the opinion of the investigator.
* Subject has completed the ACSM exercise preparticipation health screening and is, in the opinion of the investigator, fit to participate in this study.

Exclusion Criteria:

-Currently adhering to national physical activity guidelines for resistance training, as defined as participating in structured resistance training ≥ two days per week.

* Structured is defined as time set aside in the subject's day to workout.
* Resistance training is defined as exercises which use weights, bands, or body weight (e.g., squats or push-ups).

AND Currently participating in structured moderate-intensity aerobic exercise for ≥ 150 minutes per week.

* Moderate-intensity exercise is defined as activities where the subject can talk but not sing.
* Aerobic exercise includes, but is not limited to, walking, swimming, cycling, running, rowing, hiking, and elliptical.

  * Medical, psychiatric, cognitive, or other conditions that may compromise the participant's ability to understand the participant information, give informed consent, comply with the study protocol or complete the study.
  * Participants taking prohibited medications as described in Section 6.4.1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-11-04 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Change in Functional Assessment of Chronic Illness Therapy (FACIT) Fatigue score from baseline to Week 13 (end of exercise intervention). | 13 weeks
  Test the preliminary efficacy of a 12-week, home-based, unsupervised aerobic and resistance training exercise program on changes in cancer-related fatigue, in patients with Metastatic Breast Cancer recently initiated on Enhertu. FACIT Fatigue Scored 0 (not at all)- 4(Very Much).

SECONDARY OUTCOMES:
Feasibility defined as greater than 75% of all participants completing greater than 66% of all prescribed workouts from baseline to Week 13. | 13 weeks
  Test the feasibility of the tested 12-week, home-based, unsupervised aerobic and resistance training exercise program.
Mean Functional Assessment of Chronic Illness Therapy (FACIT) Fatigue score measured every three weeks from baseline to Week 13. | 13 weeks
  Compare the trajectory of cancer-related fatigue from baseline to Week 13 between patients receiving the exercise intervention versus not. FACIT Fatigue Scored 0 (not at all)- 4 (Very Much).

OTHER OUTCOMES:
Change in Functional Assessment of Cancer Therapy - Breast (FACT-B) score from baseline to Week 13. | 13 weeks
  Evaluate the preliminary efficacy of the exercise intervention on breast cancer-related quality of life. FACT-B scored 0 (not at all)- 4 (Very Much).
Mean Functional Assessment of Cancer Therapy - Breast (FACT-B) score measured every three weeks from baseline to 13 weeks after initiation of training. | 13 weeks
  Compare the trajectory of breast cancer-related quality of life from baseline to Week 13 after initiation of training between patients receiving the exercise intervention versus not. FACT-B scored 0 (not at all)- 4 (Very Much).
Change in the average time spent in moderate to vigorous physical activity (in minutes) | 12 weeks
  Evaluate the preliminary efficacy of the exercise intervention on exercise engagement. At one week prior to baseline (i.e. baseline), at the midpoint of the intervention (Week 6) and during the final week of the intervention (Week 12), as measured by the Actigraph GT9x Link accelerometer.
Markers evaluating activity collected from the Actigraph, such as time spent in light activity. | 12 weeks
  Evaluate the preliminary efficacy of the exercise intervention on exercise engagement.
Markers evaluating activity collected from the Actigraph, such as step count. | 12 weeks
  Evaluate the preliminary efficacy of the exercise intervention on exercise engagement.
Average time spent in moderate to vigorous physical activity (in minutes) measured at baseline, Week 6, and Week 12 by the Actigraph GT9x Link accelerometer. | 12 weeks
  Compare the trajectory of exercise engagement from baseline to 12 weeks between patients receiving the exercise intervention versus not.
Other markers evaluating activity collected daily from the Actigraph GT9x, such as step count. | 12 weeks
  Compare the trajectory of exercise engagement from baseline to 12 weeks between patients receiving the exercise intervention versus not.
Other markers evaluating activity collected daily from the Actigraph GT9x, such as time spent in light activity. | 12 weeks
  Compare the trajectory of exercise engagement from baseline to 12 weeks between patients receiving the exercise intervention versus not.
Change in mean PROMIS Physical Function score from baseline to Week 13. | 13 weeks
  Evaluate the preliminary efficacy of the exercise intervention on physical function. Scored 5 (Without any difficulty)- 1 (Unable to do).
Change in the following objective measures of physical function from baseline to Week 13: 30-second chair stand. | 13 weeks
  Evaluate the preliminary efficacy of the exercise intervention on physical function.
Change in the following objective measures of physical function from baseline to Week 13: Balance Test | 13 weeks
  Evaluate the preliminary efficacy of the exercise intervention on physical function. The Balance Test will consist of: Participants will be instructed to stand up with their feet in three different positions (side-by-side, tandem and semi-tandem) for 10 seconds each position.
Change in the following objective measures of physical function from baseline to Week 13: 30-second maximum push-up test. | 13 weeks
  Evaluate the preliminary efficacy of the exercise intervention on physical function.
Average physical function measured at baseline, Week 6, and Week 12 by PROMIS Physical Function score. | 12 weeks
  Compare the trajectory of physical function from baseline to 12 weeks between patients receiving the exercise intervention versus not. Scored 5 (Without any difficulty)- 1 (Unable to do).
Other markers evaluating physical function, including 30-second chair stand. | 12 weeks.
  Compare the trajectory of physical function from baseline to 12 weeks between patients receiving the exercise intervention versus not.
Other markers evaluating physical function, including a Balance Test. | 12 weeks.
  Compare the trajectory of physical function from baseline to 12 weeks between patients receiving the exercise intervention versus not.
  The Balance Test will consist of: Participants will be instructed to stand up with their feet in three different positions (side-by-side, tandem and semi-tandem) for 10 seconds each position.
Other markers evaluating physical function, including a 30-second maximum push-up test. | 12 weeks.
  Compare the trajectory of physical function from baseline to 12 weeks between patients receiving the exercise intervention versus not.
Change in Sit-to-Stand score patterns as measured by actigraphy (central measure of fatigue) from baseline to Week 13. | 13 weeks
  Evaluate the preliminary efficacy of the exercise intervention on measures of peripheral and central fatigue.
Change in handgrip strength (peripheral measures of fatigue) patterns as measured by actigraphy (central measure of fatigue) from baseline to Week 13. | 13 weeks
  Evaluate the preliminary efficacy of the exercise intervention on measures of peripheral and central fatigue.
Change in the number of rest-activity patterns as measured by actigraphy (central measure of fatigue) from baseline to Week 13. | 13 weeks
  Evaluate the preliminary efficacy of the exercise intervention on measures of peripheral and central fatigue.
Mean score for sit-to-stand patterns measured at baseline, 6-weeks, and Week 13. | 13 weeks
  Compare the trajectory of measures of peripheral and central fatigue baseline to Week 13 after initiation of training between patients receiving the exercise intervention versus not.
Mean score for handgrip strength patterns measured at baseline, 6-weeks, and Week 13. | 13 weeks
  Compare the trajectory of measures of peripheral and central fatigue baseline to Week 13 after initiation of training between patients receiving the exercise intervention versus not.
Mean number of rest-activity patterns measured at baseline, 6-weeks, and Week 13. | 13 weeks
  Compare the trajectory of measures of peripheral and central fatigue baseline to Week 13 after initiation of training between patients receiving the exercise intervention versus not.

CONTACTS AND LOCATIONS:
Locations (1):
- Huntsman Cancer Institute at University of Utah, Salt Lake City, Utah, United States